CLINICAL TRIAL: NCT04737720
Title: Analysis of Samples Collected From a Subject Who Received ACP- 501 (Human Recombinant Lecithin:Cholesterol Acyltransferase [rhLCAT])
Brief Title: Intravenous ACP-501 for Familial LCAT Deficiency (rhLCAT)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130060; 13-H-0060
Record Dates: First submitted 2021-02-03; First posted 2021-02-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09-22

CONDITIONS: Familial LCAT Deficiency
Keywords: Recombinant LCAT; Natural History
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This is an expanded use protocol for a named subject.
  Interventions: Drug: Recombinant LCAT

INTERVENTIONS:
Drug: Recombinant LCAT — iv infusion

SUMMARY:
Background:

* High density lipoprotein (HDL), or good cholesterol, moves cholesterol from the artery walls back to the liver. A blood enzyme known as LCAT maintains HDL levels and helps it remove cholesterol from the body. Familial LCAT deficiency (FLD) is a genetic disease that results in low levels or total absence of LCAT. People with FLD often have kidney problems, and may develop kidney failure. Researchers think that the clinical problems of FLD can be prevented or even reversed by replacing the defective enzyme.
* There are no drugs that increase LCAT. It has to be artificially made and infused into the body. The artificial LCAT is called recombinant human LCAT, or ACP-501. Researchers want to see how well it works in one person with FLD and poor kidney function.

Objectives:

- To see whether ACP-501 can improve the symptoms of FLD.

Eligibility:

- One person (the study participant) with FLD.

Design:

* The participant will be screened with a physical exam and medical history. Blood samples will be collected.
* The participant will receive ACP-501 and remain in the hospital for 24 hours for regular blood tests. The participant may stay in the hospital or return for daily clinic visits until it is time for the next dose. The second dose will be given on Day 4 or Day 8.
* If an optimal dose has not yet been identified, a third dose will be given 7 days after the second dose.
* The participant will then go home, but must return to the hospital for ACP-501 infusions and blood tests every 1 or 2 weeks, as needed. Every 3 months, the participant will have a full clinic visit with blood tests and other studies.

DETAILED DESCRIPTION:
This primary objective of the study was to use ACP-501 (recombinant LCAT - rhLCAT) as an Expanded Access Protocol in order for one named subject with Familial LCAT Deficiency (FLD) with the hope of slowing or preventing the progression of renal dysfunction and eliminating the need for dialysis. This was a first-in-human study of ACP-501 (rhLCAT) in a subject with FLD. The safety and tolerability of rhLCAT, was assessed after multiple infusions. The pharmacokinetics (PK) of rhLCAT and its effect on the pharmacodynamics (PD) of HDL-C and HDL subpopulations was also be assessed. The duration of the PK and PD parameters will inform future multiple dose studies with respect to dose (mg/kg) and dosing interval. The current protocol completed the primary objection and has shifted to the secondary analysis of samples that were collected. FLD is an extremely rare generic disorders and there are too few subjects to design additional phase 1 trials and these longitudinal samples demonstrating the appearance of normal HDL along with possible biomarkers will be helpful and can help guide the design of a small definitive phase II/II trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Greater than or equal to 18 years at screening;
* Confirmed FLD diagnosis through genotype confirmation of a LCAT mutation, as documented at screening or from previous testing;
* History of HDL-C < 15 mg/dL over the past year;
* Serum creatinine > 3 mg/dL;
* Increasing renal dysfunction resulting in ESRD;
* Chronic concomitant medications must be stable for at least 2 weeks prior to screening (for example, lipid-altering drugs and/or ACE-inhibitors used for the treatment of FLD).
* Subject is willing and able to comply with scheduled study visits and is able to tolerate study procedures, including weekly to bi-weekly infusions over 1 year.
* Subject must be able to provide a personally-signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subject may be currently on dialysis or require dialysis during the study

EXCLUSION CRITERIA:

Subject will not be included in the study if he presents with any of the following:

* History of febrile illness within 5 days prior to dosing;
* Active non-basal cell cutaneous malignancy requiring surgery, chemotherapy, and/or radiation in the past 12 months.

NOTE: Subjects with localized prostate cancer under a watchful-waiting treatment plan without evidence of disease progression in the past year may participate in the study if approved by the investigator and sponsor or designee.

NOTE: Subjects diagnosed with basal cell carcinoma of the skin within the past 12 months must receive adequate treatment for their basal cell skin carcinoma prior to randomization.

* Current documented drug or alcohol abuse that would interfere with the subject s compliance with study procedures;
* Treatment with an investigational drug within 28 days prior to dosing.
* Known hypersensitivity to heparin or IV infusion equipment, plastics, adhesive or silicone or known history of hypotension or infusion site reactions with IV administration.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial or compromise the subject s ability to continue with the procedures of the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2013-12-12 (Actual)

PRIMARY OUTCOMES:
HDL | weekly
  Increased

SECONDARY OUTCOMES:
LCAT | weekly
  Increased

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a single patient expanded access study.

REFERENCES:
- [Background] Barter PJ. Hugh sinclair lecture: the regulation and remodelling of HDL by plasma factors. Atheroscler Suppl. 2002 Dec;3(4):39-47. doi: 10.1016/s1567-5688(02)00041-7. PMID 12573362
- [Background] Lee JY, Badeau RM, Mulya A, Boudyguina E, Gebre AK, Smith TL, Parks JS. Functional LCAT deficiency in human apolipoprotein A-I transgenic, SR-BI knockout mice. J Lipid Res. 2007 May;48(5):1052-61. doi: 10.1194/jlr.M600417-JLR200. Epub 2007 Feb 1. PMID 17272829
- [Background] Rousset X, Vaisman B, Amar M, Sethi AA, Remaley AT. Lecithin: cholesterol acyltransferase--from biochemistry to role in cardiovascular disease. Curr Opin Endocrinol Diabetes Obes. 2009 Apr;16(2):163-71. doi: 10.1097/med.0b013e328329233b. PMID 19306528
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0060.html